CLINICAL TRIAL: NCT00693498
Title: Standard vs. Washed Blood Cell Transfusions in Pediatric Cardiac Surgery: Impact on Post-operative Inflammation as Evidenced by the IL-6 to IL-10 Ratio.
Brief Title: Washed Versus Standard Blood Cell Transfusions in Pediatric Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jill Cholette, Assistant Professior, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24518
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Results first posted 2012-11-29 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Congenital Heart Disease
Keywords: pediatrics; congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Standard leukoreduced irradiated blood cell transfusion group
  Interventions: Biological: Standard leukoreduced irradiated blood cell transfusion
- 2 (Experimental): Washed leukoreduced irradiated blood cell transfusion group
  Interventions: Biological: Washed leukoreduced irradiated blood cell transfusions

INTERVENTIONS:
Biological: Standard leukoreduced irradiated blood cell transfusion — standard vs washed blood cell transfusions
  Arms: 1
Biological: Washed leukoreduced irradiated blood cell transfusions — washed leukoreduced irradiated blood cell transfusions
  Arms: 2

SUMMARY:
Background: Children having open heart surgery to repair congenital heart defects demonstrate a large inflammatory response to the heart-lung machine and to surgery itself. In general, the more intense their inflammatory response, the more critically ill they are following surgery. These children routinely require large numbers of blood transfusions during and following surgery as part of their medical management that adds to their heightened inflammatory state. Whether additional steps to "wash" blood products and remove the substances contributing to post-transfusion inflammation will limit this response, and improve the health of children following open heart surgery, remains to be studied.

Aims: To compare the inflammatory response in children having open heart surgery who receive washed versus unwashed blood transfusions.

Methods: We will randomly assign children having open heart surgery to one of two groups: group 1 will receive blood transfusions per the current standard of care, group 2 will receive blood transfusions that have been washed in addition to the current standard of care. We will then use blood tests to measure the inflammatory response in children of each group. We will compare the results to determine whether washing blood transfusions decreases inflammation and post-operative complications following open heart surgery.

Conclusion: We believe that washing blood transfusions given to children following open heart surgery will decrease their inflammatory response and improve their overall health.

ELIGIBILITY:
Inclusion Criteria:

1. age < 18 years
2. surgical repair at URMC by the pediatric cardiac surgical team
3. informed consent signed by the parent or legal guardian, and if applicable, assent obtained from the subject.

Exclusion Criteria:

1. Age ≥18 years
2. inability to provide consent/assent; 3) subjects having "emergent" surgical procedures. Subjects with chronic inflammatory or autoimmune disorders will not be excluded

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2008-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Cholette, MD, Principal Investigator — University of Rochester

REFERENCES:
- [Derived] Cholette JM, Henrichs KF, Alfieris GM, Powers KS, Phipps R, Spinelli SL, Swartz M, Gensini F, Daugherty LE, Nazarian E, Rubenstein JS, Sweeney D, Eaton M, Lerner NB, Blumberg N. Washing red blood cells and platelets transfused in cardiac surgery reduces postoperative inflammation and number of transfusions: results of a prospective, randomized, controlled clinical trial. Pediatr Crit Care Med. 2012 May;13(3):290-9. doi: 10.1097/PCC.0b013e31822f173c. PMID 21926663

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects were recruited at pre-anesthesia inpatient assessments and outpatient pre-anesthesia appointments.
Groups:
- Standard Transfusion Group: Standard leukoreduced irradiated ABO compatible red blood cell and platelet transfusion group
- Washed Transfusion Group: Washed leukoreduced irradiated ABO compatible red blood cell and platelet transfusion group
Period: Overall Study
Arm/Group | Standard Transfusion Group | Washed Transfusion Group
Started | 81 | 81
Completed | 81 | 81
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Transfusion Group | Washed Transfusion Group | Total
Number analyzed (Participants) | 81 | 81 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 81 | 81 | 162
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: days]
  Age | 1 (NA) [1 to 17] | 1 [1 to 17] | 1 [1 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 64 | 63 | 127

OUTCOME MEASURES:

1. Primary Outcome: 12 Hour Plasma Interleukin (IL)-6 to IL-10 Ratio
Description: plasma was obtained pre-op, immediately once off cardiopulmonary bypass (CPB), six hours following CPB and 12 hours following CPB. The plasma was centrifuged and the supernatant collected and stored at -70 degrees. The samples then underwent Luminex testing for IL-6 and IL-10 levels, and the IL-6:IL-10 ratio was calculated (IL-6 being the numerator and IL-12 being the denominator). The 12 hour ratio was the primary outcome measure.
Time Frame: 12 hours post-cardiopulmonary bypass
Population: Only data from those subjects receiving transfusions was analyzed as the study intervention was the type of red blood cell and platelet transfusion (washed v. unwashed).
Measure: Median (Standard Error); unit: ratio
Arm/Group | Standard Transfusion Group | Washed Transfusion Group
Number analyzed (Participants) | 64 | 64
ratio | 8.9 (1.2) | 3.8 (1.3)

2. Secondary Outcome: Median wrCRP Level
Description: wide range C reactive protein levels were obtained before surgery (pre-operatively) and on post-operative day 1 and 2 in transfused subjects
Time Frame: post op day 1 and 2
Population: 64 subjects in each group that received blood; all included in the analysis
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Standard Transfusion Group | Washed Transfusion Group
Number analyzed (Participants) | 64 | 64
mg/dL
  POD #1 | 43 [0 to 300] | 38 [0 to 85]
  POD #2 | 70 [0 to 375] | 59 [0 to 175]
Statistical Analysis 1: Comparison: Standard Transfusion Group vs Washed Transfusion Group; Test type: Other; p < 0.03, Wald Wolfowitz — the reported value is for POD#1 assessment
Statistical Analysis 2: Comparison: Standard Transfusion Group vs Washed Transfusion Group; Test type: Other; p = 0.29, Wald-Wolf — for POD#2 assessment

ADVERSE EVENTS:
Arm/Group | Standard Transfusion Group | Washed Transfusion Group
Serious Adverse Events (participants affected / at risk) | 6/81 | 2/81
Other Adverse Events (participants affected / at risk) | 13/81 | 13/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Transfusion Group (N=81) | Washed Transfusion Group (N=81)
Death (Cardiac disorders) | 6 (6) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Transfusion Group (N=81) | Washed Transfusion Group (N=81)
Infection (Infections and infestations) | 13 (13) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No